CLINICAL TRIAL: NCT04372303
Title: Effect of a Compassion Fatigue Resiliency Program on Nurses' Professional Quality of Life, Perceived Stress, Resilience: A Randomized Controlled Trial
Brief Title: Effect of a Compassion Fatigue Resiliency Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Pehlivan, Principal Investigator, Koc University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TPehlivan
Record Dates: First submitted 2020-04-23; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Compassion Fatigue
Keywords: Oncology-hematology nurses; compassion fatigue; burnout; compassion satisfaction; perceived stress; resilience
MeSH Terms: conditions — Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short-term Compassion Fatigue Resiliency Program (Experimental): Experimental I received a short-term program (five hours per day for two days, ten hours in total).
  Interventions: Behavioral: Compassion Fatigue Resiliency Program (CFRP)
- Long-term Compassion Fatigue Resiliency Program (Experimental): Experimental II received a long-term program (five weeks, two hours per week, ten hours in total).
  Interventions: Behavioral: Compassion Fatigue Resiliency Program (CFRP)
- Control (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Behavioral: Compassion Fatigue Resiliency Program (CFRP) — The purpose of Compassion Fatigue Resiliency Program (CFRP) is to provide oncology-hematology nurses with knowledge and skills that will increase their level of resilience by helping them recognize compassion fatigue, cope with its consequences and work effectively.
  Arms: Long-term Compassion Fatigue Resiliency Program; Short-term Compassion Fatigue Resiliency Program

SUMMARY:
This study aimed to conduct a short- and long-term Compassion Fatigue Resiliency Program and compare its impact on nurses' professional quality of life, perceived stress and resilience. The research was conducted between January 2017 and January 2019 as a randomized controlled trial. The sample comprised 125 oncology-hematology nurses randomly assigned to a Experimental I (short-term Compassion Fatigue Resiliency Program), Experimental II (long-term Compassion Fatigue Resiliency Program) or control group. Data was collected using Personal Information Form, Professional Quality of Life Scale-IV (ProQOL-IV), Perceived Stress Scale, and Resilience Scale for Adults. Measurements were obtained during pre- and post-test and at three-, six- and twelve-month follow-ups. Research hypotheses were analyzed using multilevel models.

DETAILED DESCRIPTION:
The research was conducted with nurses from the oncology-hematology inpatient services, outpatient chemotherapy units and bone marrow transplant (BMT) units of three private hospitals in Istanbul between January 2017 and January 2019. No sample selection models were applied, and out of 153 nurses working in these services, 125 nurses meeting the inclusion criteria were included in the study. Nurses were randomly assigned to the Experimental I, Experimental II, or control group in order to prevent interaction between the subjects working in the same hospital. Of the nurses, 34 completed the short-term program (Experimental I), 49 completed the long-term (Experimental II), and 42 were assigned to the control group.

Data collection: Data was collected using Personal Information Form, Professional Quality of Life Scale-IV (ProQOL-IV), Perceived Stress Scale, and Resilience Scale for Adults Study procedure This study's principal investigator had participated online in a CFRP, developed by Eric Gentry (Licensed Mental Health Counselor) (2002), and received the certificate, and then conducted the program with the nurses. Meetings were held with each institution's directorate of nursing services to determine the training schedules and content. The schedules were planned in accordance with the hospital administration's preferences and by taking nurses' busy schedules into consideration. Preliminary tests were applied to Experimental I, Experiment II, and the control group before the training. Experimental I received a short-term program (five hours per day for two days, ten hours in total) while Experimental II received a long-term one (five weeks, two hours per week, ten hours in total). No intervention was applied to the control group. After the training, a post-test, and three-, six-, and twelve-month follow-up assessments were conducted for all groups.

Program Compassion Fatigue Resiliency Program The purpose of the program: The purpose of the program is to provide oncology-hematology nurses with knowledge and skills that will increase their level of resilience by helping them recognize compassion fatigue, cope with its consequences and work effectively.

The objectives of the training program

Nurses, who successfully complete the program will be able to:

* Explain the historical development of compassion fatigue among caregivers,
* Define the developmental process of compassion fatigue,
* Specify the risk factors for compassion fatigue,
* Explain the symptoms of compassion fatigue,
* Raise awareness about their personal history,
* Explain the concept of stress and its impact on the body,
* Apply compassion fatigue resilience skills acquired in the program,
* Professionally create a self-directed resilience plan. Validity and reliability/Rigour The included scales have been tested for validity and reliability for various settings and countries. The investigators chose three private hospitals in Istanbul, which are considered to be close to each other, such as institution (etc. working conditions) and the sociodemographic and professional characteristics of nurses (etc. age, educational status, clinical experience, willingness to work in oncology, voluntarily career choice) that are known to affect dependent variables. Then, the investigators randomly assigned each hospital to the Experimental I, Experimental II, or control group in order to prevent interaction between the nurses working in the same hospital. Finally, the program was conducted by the principal investigator who had participated online in a CFRP, and received the certificate.

Data analysis: SPSS 25.0 software package was used to analyze data. A chi-square test and one-way ANOVA determined whether the scales and information on demographic characteristics and work environment differed among pre-initiative groups; in other words, to measure homogeneity. Variables found to be statistically significant were included in the model as a correction factor for primary hypotheses. Primary research hypotheses were analyzed using multilevel models (MLM). This analysis method has some advantages over others, such as repeated measures ANOVA.

ELIGIBILITY:
Inclusion criteria

* Nurses working in inpatient oncology-hematology, outpatient chemotherapy, or BMT unit Exclusion criteria
* Providing care for pediatric oncology patients
* Being a nurse manager
* Not providing direct patient care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Professional Quality of Life Scale-IV (ProQoL), "change" is being assessed. | Change from Baseline up to 1 year
  Professional Quality of Life Scale-IV (ProQoL): It is a self-reporting instrument consisting of thirty items and three subscales: Compassion Fatigue (CF), Sompassion Satisfaction (CS), and burnout. The scale has no total score. Each subscale is evaluated separately.
  * Scores above 17 indicate high CF levels while scores below 8 indicate low,
  * Scores below 18 indicate low burnout levels while scores above 27 indicate high
  * Scores above 42 indicate high CS levels while those below 33 indicate low
Perceived Stress Scale, "change" is being assessed. | Change from Baseline up to 1 year
  Perceived Stress Scale: The lowest possible score is 0 and the highest is 40. A high total score is considered a high level of perceived stress.
Resilience Scale for Adults, "change" is being assessed. | Change from Baseline up to 1 year
  Resilience Scale for Adults: a lowest possible score of 33 and a highest of 165. A high total score is considered a high level of resilience.

IPD SHARING:
Plan to Share IPD: No
No, because hospitals told us, the investigators have to keep secret their nurses individual data.

REFERENCES:
- [Background] Traeger L, Park ER, Sporn N, Repper-DeLisi J, Convery MS, Jacobo M, Pirl WF. Development and evaluation of targeted psychological skills training for oncology nurses in managing stressful patient and family encounters. Oncol Nurs Forum. 2013 Jul;40(4):E327-36. doi: 10.1188/13.ONF.E327-E336. PMID 23803277
- [Background] Tarantino B, Earley M, Audia D, D'Adamo C, Berman B. Qualitative and quantitative evaluation of a pilot integrative coping and resiliency program for healthcare professionals. Explore (NY). 2013 Jan-Feb;9(1):44-7. doi: 10.1016/j.explore.2012.10.002. PMID 23294820
- [Background] Deible S, Fioravanti M, Tarantino B, Cohen S. Implementation of an integrative coping and resiliency program for nurses. Glob Adv Health Med. 2015 Jan;4(1):28-33. doi: 10.7453/gahmj.2014.057. PMID 25694849
- [Background] Rushton CH, Batcheller J, Schroeder K, Donohue P. Burnout and Resilience Among Nurses Practicing in High-Intensity Settings. Am J Crit Care. 2015 Sep;24(5):412-20. doi: 10.4037/ajcc2015291. PMID 26330434
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Friborg O, Barlaug D, Martinussen M, Rosenvinge JH, Hjemdal O. Resilience in relation to personality and intelligence. Int J Methods Psychiatr Res. 2005;14(1):29-42. doi: 10.1002/mpr.15. PMID 16097398
- [Derived] Pehlivan T, Guner P. Effect of a compassion fatigue resiliency program on nurses' professional quality of life, perceived stress, resilience: A randomized controlled trial. J Adv Nurs. 2020 Dec;76(12):3584-3596. doi: 10.1111/jan.14568. Epub 2020 Oct 3. PMID 33009840
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860